CLINICAL TRIAL: NCT03464786
Title: A Clinical Study on the Efficacy and Safety of Lando® Absorbable Collagen Membrane in Oral Bone Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Lando Biomaterials Co., Ltd. (Industry)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LD-M-201701
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- absorbable collagen membrane (Experimental): Subjects randomized in this arm will receive Lando® absorbable collagen membrane after tooth extraction.
  Interventions: Device: Lando® absorbable collagen membrane
- Bio-Gide resorbable bilayer membrane (Active Comparator): Subjects randomized in this arm will receive Bio-Gide resorbable bilayer membrane after tooth extraction.
  Interventions: Device: Geistlich Bio-Gide resorbable bilayer membrane

INTERVENTIONS:
Device: Lando® absorbable collagen membrane — Subjects who are fit for the study will be randomized to either intervention arms.
  Arms: absorbable collagen membrane
Device: Geistlich Bio-Gide resorbable bilayer membrane — Subjects who are fit for the study will be randomized to either intervention arms.
  Arms: Bio-Gide resorbable bilayer membrane

SUMMARY:
This is a randomized, paralleled, control trial to validate the effectiveness and safety of Lando® absorbable collagen membrane for oral bone repair.

ELIGIBILITY:
Inclusion Criteria:

* 18~65 years old;
* Subjects, whose single teeth (adjacent teeth intact) of incisor, canine or premolar is removed and bone graft is needed for alveolar ridge preservation, and need a delayed implant repair in more than 26 weeks.
* voluntary participation and sign on the informed consent form

Exclusion Criteria:

* Participated in other clinical trials in 90 days before joined in the trial
* Having received in 90 days before joined in the trial and / or will receive the head and neck radiation therapy or chemist during the study
* Having received in 90 days before joined in the trial and / or will receive any drug treatment that may affect bone metabolism;
* patients with heart disease;
* patients with abnormal liver and kidney function;
* poor diabetes control;
* low or abnormal immunity, anaphylaxis and the researchers judged to be of clinical significance;
* HIV infected patients;
* bleeding tendency or coagulation disorders and researchers judged to be of clinical significance;
* mental disorder;
* women who are pregnant or breast-feeding or preparing for pregnancy in the next 26 weeks;
* severe smokers;
* patients with periodontitis without basic periodontal treatment;
* the fracture of alveolar process after tooth extraction;
* The loss of bone wall on any side of alveolar fossa was more than 2/3.
* other cases that researchers believe not suitable for the participants of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Change value of the width of alveolar ridge | 26 weeks
  Change value of the width of alveolar ridge by CT

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Stomatological Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No